CLINICAL TRIAL: NCT02187588
Title: Short Term Double Blind Randomised Controlled Study to Assess the Kinetic of the Analgesic Effect and the Tolerability of Eschscholtzia Californica 500 mg and 1000 mg Versus Ibuprofen 200 mg and Placebo in the Treatment of Pain After Surgery of the Third Molar
Brief Title: Study to Assess the Kinetic of the Analgesic Effect and Tolerability of Eschscholtzia Californica Versus Ibuprofen and Placebo in the Treatment of Pain After Surgery of the Third Molar
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1120.3
Record Dates: First submitted 2014-07-10; First posted 2014-07-11 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Ibuprofen

ARMS (4):
- Eschscholtzia Californica - low dose (Experimental)
  Interventions: Drug: Eschscholtzia Californica - low dose; Drug: Eschscholtzia Californica - low dose Placebo; Drug: Ibuprofen Placebo
- Eschscholtzia Californica - high dose (Experimental)
  Interventions: Drug: Eschscholtzia Californica - high dose; Drug: Ibuprofen Placebo
- Ibuprofen (Active Comparator)
  Interventions: Drug: Ibuprofen; Drug: Eschscholtzia Californica - high dose Placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: Eschscholtzia Californica - high dose Placebo; Drug: Ibuprofen Placebo

INTERVENTIONS:
Drug: Eschscholtzia Californica - low dose
  Arms: Eschscholtzia Californica - low dose
Drug: Eschscholtzia Californica - high dose
  Arms: Eschscholtzia Californica - high dose
Drug: Ibuprofen
  Arms: Ibuprofen
Drug: Eschscholtzia Californica - low dose Placebo
  Arms: Eschscholtzia Californica - low dose
Drug: Eschscholtzia Californica - high dose Placebo
  Arms: Ibuprofen; Placebo
Drug: Ibuprofen Placebo
  Arms: Eschscholtzia Californica - high dose; Eschscholtzia Californica - low dose; Placebo

SUMMARY:
Study to determine the kinetic of the analgesic effect of 500 mg and 1000 mg of Eschscholtzia Californica per os and placebo in patients undergoing dental surgery over an observation period of 6 hours. In a secondary analysis, kinetic of analgesic effect comparison between Eschscholtzia californica 500 mg, 1000 mg and Ibuprofen 200 mg

ELIGIBILITY:
Inclusion Criteria:

* Male or female above 18 or below 61 years old
* Patient having to undergo a third molar removal from the lower jaw under local troncular anesthesia (articaine + adrenaline)
* Type of inclusion of the molar:

  * Molar in the sub-mucosa: Type II
  * Molar partially impacted in the bone: Type III
* Patient suffering from at least moderate to severe pain after surgical removal of an impacted third molar, defined by a 4 point verbal rating scale
* Patient's informed consent in accordance with the French legislation
* Patient affiliated to the Social Security System

Exclusion Criteria:

* Pregnant or nursing female or female of childbearing potential not using a medically approved method of contraception like oral contraception or intrauterine contraceptive device
* Patient with any pathology inducing a chronic pain
* Patient having taken any drug with analgesic properties in the 24 hours previous to the administration of the study drug
* Patient with concomitant administration of other Non-Steroid Anti-Inflammatory Drug(s) (NSAIDs) or analgesic agents
* Patients treated by an antibiotic different from those required for the dental surgery which administration is started 48 hours prior to the tooth removal
* Patient with significant peri-operative complication judged by the investigator
* Patient with anti-coagulants concomitant treatment (including heparin)
* Patient with severe hepatic or renal insufficiency which judged to be regarded as clinically relevant by the investigator or any known clinically significant disease which may induce a risk for the patient in participating to the trial
* Patient with mental disturbance
* Patient with non controlled diabetes
* Patient with acute infections
* Patient with respiratory insufficiency, asthma
* Patient unable to comply with the protocol
* Patient having taken part in a clinical trial in the past month or already participating in another trial
* Patient deprived of their freedom by a judicial or administrative decision
* Adults under guardianship
* Persons hospitalized in medical or social establishments
* Patients in emergency situation
* Patient with a known or suspected hypersensitivity to the trial medication, to Ibuprofen, Paracetamol, anesthetic used (articaine, adrenaline), to the preventive antibiotic treatment (penicillin, macrolides)

Post study exclusion period: the patient will not be able to participate in any other trial for a period of two weeks after the end of this trial

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 1998-02; Primary Completion 1999-05 (Actual)

PRIMARY OUTCOMES:
VAS-SPID - summed pain intensity differences (SPID) on a VAS (Visual Analogue Scale) | Baseline, up to 6 hours after drug intake

SECONDARY OUTCOMES:
Pain intensity differences (PID) on a VAS | Baseline, up to 6 hours after drug intake
Pain intensity difference in the groups on a VAS | Baseline, 2 hours after drug intake
Time point for maximum pain intensity difference on VAS | Baseline, up to 6 hours after drug intake
Number of patients with a pain decrease of at least 50 % over the all period of observation on a VAS | Baseline, up to 6 hours after drug intake
Pain relief at each observed time points on a 5-point verbal rating scale (VRS) | up to 6 hours after drug intake
Total pain relief on a 5-point VRS | up to 6 hours after drug intake
Global efficacy assessment on a 4-points VRS | 2 and 6 hours after drug intake, day 7
Number of patients requiring a rescue medication | Day 1
Number of patients with adverse events | up to 9 days after treatment
Assessment of tolerability by investigator on a 4-point VRS | 6 hours after drug intake, day 7
Assessment of tolerability by subject on a 4-point VRS | 6 hours after drug intake, day 7